CLINICAL TRIAL: NCT03266432
Title: Thromboelastometry Guided Disseminated Intravascular Coagulation Prevention After Cesarean Section in Pregnant Women With Placenta Previa
Brief Title: Thromboelastometry Guided DIC Prevention After Cesarean Section in Pregnant Women With Placenta Previa
Acronym: DIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Kilany, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: thromboelastometryDIC
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: DIC Syndrome
MeSH Terms: conditions — Disseminated Intravascular Coagulation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 60 pregnant women (Other): 60 pregnant women diagnosed with placenta previa will take from them 3 blood samples : one pre intervention and two samples postintervention
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — three blood samples : first one pre intervention and the other two blood samples post-intervention

SUMMARY:
Evaluation of the use of thromboelastometry for early identification of the underlying coagulopathy and to guide individualized transfusion therapy to prevent DIC development during ICU stay after cesarean section in women with placenta previa who require a massive blood transfusion.

DETAILED DESCRIPTION:
Placenta previa is defined as complete or partial implantation of the placenta in the lower segment of the uterus, Patients present with bleeding per vagina occurring usually in the second and third trimester. Bleeding in placenta previa is associated with maternal morbidity and mortality. Transfusion therapy is integral in the acute management of major obstetric hemorrhage. The most important pregnancy related condition leading to bleeding with high mortality and morbidity rates is DIC. Patients exhibit a tendency for severe bleeding associated with the consumption of platelets and coagulation factors. Massive blood transfusions are listed as the main maternal morbidity indicators6.Therefore, early detection of these predictors of DIC and timely intervention of this life-threatening condition is very important. DIC is a clinical-laboratory diagnosis, and laboratory changes need to be interpreted with knowledge of the patient's underlying disorder. Several laboratory parameters are analyzed together as part of a diagnostic algorithm that includes: Prothrombin time (PT), Activated partial thromboplastin time (aPTT), the platelet count, fibrinogen level, and a marker of fibrin degradation, e.g., D-dimer or the soluble fibrin monomer (SFM) 8. None of these markers are taken in isolation, and a combination of results at different time points is particularly helpful in determining the presence of DIC, owing to the multifaceted nature of DIC9, These reasons highlight a strong need for the development of a point-of-care testing system to accurately and reliably diagnose DIC. Thromboelastography (TEM) provides an extended reflection of clot initiation, propagation, and lysis in whole blood. TEM uses three tests: FIBTEM to reveal impaired fibrinogen function, INTEM to reveal coagulation factor deficiency and EXTEM to reveal extrinsic pathway defects

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Age: ≥ 18 years
* Patients with all types of placenta previa
* Eligible for general anesthesia
* Elective cesarean section
* Singleton term pregnancy
* Normal coagulation profile: prothrombin time (PT), activated partial thromboplastin time (aPTT), the platelet count, fibrinogen level

Exclusion Criteria:

* Parturient refusal
* Known coagulopathy
* Women with a history of cardiac, respiratory, renal, neurologic or endocrine diseases.
* Eclampsia and preeclampsia
* Emergency surgeries
* Foetal abnormalities
* Drug induced thrombocytopenia as antibiotics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
prevention of Postoperative development of DIC | from time of operation till 48 hours postopertive
  prevention according to the results of thromboelastometry

SECONDARY OUTCOMES:
prevention of Complications of massive transfusion | from time of operation till 48 hours postoperative
  hypo or hyperkalaemia, hypoc alcaemia, hypothermia and metabolic alkalosis and Length of ICU and hospital stay and In-hospital mortality
Systolic blood pressure | from time of operation till 48 hours postoperative
  systolic blood pressure is measured every hour from time of operation till 48 hours postoperative
diastolic blood pressure | from time of operation till 48 hours postoperative
  diastolic blood pressure is measured every hour from time of operation till 48 hours postoperative
heart rate | from time of operation till 48 hours postoperative
  heart rate is recorded every hour from time of operation till 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: ragaa Ahmed Herdan, MD, Principal Investigator — Assiut university hopitals
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided